CLINICAL TRIAL: NCT04947254
Title: Phase II Trial of Primary Radiotherapy With Androgen Ablation With or Without Adjuvant Niraparib for Selected High-Risk Locoregional Prostate Cancer
Brief Title: Androgen Ablation Therapy With or Without Niraparib After Radiation Therapy for the Treatment of High-Risk Localized or Locally Advanced Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1039; NCI-2021-05724 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1039 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Prostate Carcinoma; Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Androgen Antagonists; apalutamide; Biopsy; niraparib; Prednisone; deltacortene; prednylidene; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Apa, ADT, XRT) (Active Comparator): PART 1 NEOADJUVANT PHASE (CYCLES 1-3): Patients receive PO QD on days 1-28, and physician's choice ADT. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  PART 2 RADIATION PHASE (CYCLES 4-6): Within 30 days of completing Part 1, patients undergo radiation therapy. Patients also receive apalutamide PO QD on days 1-28 and physician's choice ADT. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  PART 3 ADJUVANT PHASE (CYCLES 7 AND BEYOND): Patients receive apalutamide PO QD on days 1-28 and physician's choice ADT. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Antiandrogen Therapy; Drug: Apalutamide; Procedure: Biopsy; Radiation: Radiation Therapy
- Group B (Apa, ADT, XRT, AAP, niraparib) (Experimental): PART 1 NEOADJUVANT PHASE (CYCLES 1-3): Patients receive PO QD on days 1-28, and physician's choice ADT. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  PART 2 RADIATION PHASE (CYCLES 4-6): Within 30 days of completing Part 1, patients undergo radiation therapy. Patients also receive apalutamide PO QD on days 1-28 and physician's choice ADT. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  PART 3 ADJUVANT PHASE (CYCLES 7 AND BEYOND): Patients receive abiraterone acetate PO QD, prednisone PO BID, physician's choice ADT, and niraparib PO QD. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abiraterone Acetate; Drug: Antiandrogen Therapy; Drug: Apalutamide; Procedure: Biopsy; Drug: Niraparib; Drug: Prednisone; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Abiraterone Acetate — Given PO
  Other Names: CB7630; Zytiga
  Arms: Group B (Apa, ADT, XRT, AAP, niraparib)
Drug: Antiandrogen Therapy — Given ADT
  Other Names: ADT; Androgen Deprivation Therapy; Androgen Deprivation Therapy (ADT); Anti-androgen Therapy; Anti-androgen Treatment; Antiandrogen Treatment; Hormone Deprivation Therapy; Hormone-Deprivation Therapy
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; Erleada; JNJ 56021927; JNJ-56021927
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Drug: Niraparib — Given PO
  Other Names: MK-4827; MK4827
  Arms: Group B (Apa, ADT, XRT, AAP, niraparib)
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
  Arms: Group B (Apa, ADT, XRT, AAP, niraparib)
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase II trial studies the effect of androgen ablation therapy with or without niraparib after standard of care radiation therapy in treating patients with prostate cancer that has not spread to other parts of the body (localized) or that has spread to nearby tissue or lymph nodes (locally advanced). Androgen ablation therapy (also known as hormone therapy) lowers the levels of male hormones called androgens in the body. Androgens stimulate prostate cancer cells to grow. There are 2 types of androgen ablation therapy given in this study: AAP + ADT and Apa + ADT. AAP + ADT is the treatment combination of the drugs abiraterone acetate and prednisone (AAP) given with androgen deprivation therapy (ADT, also known as androgen deprivation therapy or androgen suppression medication, which is used as standard of care to lower testosterone levels in men with high risk localized or metastatic prostate cancer). Apa + ADT is the treatment combination of the drug apalutamide (Apa) given with ADT. Androgen ablation therapy with or without niraparib after radiation therapy may help to control the disease in patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the efficacy of addition of adjuvant niraparib to maximal androgen signaling ablation (AAP + ADT) versus maximal androgen signaling ablation alone (Apa + ADT) following definitive radiation therapy (XRT) for biomarker-selected men with poor histopathologic response to neoadjuvant androgen signaling ablative therapy.

SECONDARY OBJECTIVES:

I. Determine the safety and tolerability of adjuvant niraparib with androgen ablation versus androgen ablation alone following definitive XRT in the study population.

II. Determine the impact of the addition of adjuvant niraparib to maximal androgen signaling ablation (AAP + ADT) versus maximal androgen signaling ablation alone (Apa + ADT) following definitive XRT for biomarker-selected men with good and poor histopathologic response to neoadjuvant androgen signaling ablative therapy on overall survival III. Determine the impact of the niraparib + AAP + ADT and Apa+ADT treatment on eugonadal (non-castrate levels of testosterone) progression free survival.

IV. Determine the impact of favorable versus unfavorable histologic response on progression-free survival (PFS) in men who received maximal androgen signaling ablation prior to definitive radiation.

CORRELATIVE OBJECTIVE:

I. Collect and archive solid and liquid tumor samples, as well as normal blood samples for germline deoxyribonucleic acid (DNA), immune, and metabolic profiles from all study patients for later hypothesis generating associations. Assess the relationship of histopathologic score with circulating markers and clinical outcomes of progression free survival for biomarker discovery.

OUTLINE:

PART 1 NEOADJUVANT PHASE (CYCLES 1-3): Patients receive apalutamide orally (PO) once daily (QD) on days 1-28, and physician's choice ADT. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

PART 2 RADIATION PHASE (CYCLES 4-6): Within 30 days of completing Part 1, patients undergo radiation therapy. Patients also receive apalutamide PO QD on days 1-28 and physician's choice ADT. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

PART 3 ADJUVANT PHASE (CYCLES 7 AND BEYOND): Patients with favorable response after Part 2 continue Apa + ADT. Patients with unfavorable response after Part 2 are randomized to 1 of 2 groups.

GROUP A: Patients receive apalutamide PO QD on days 1-28 and physician's choice ADT. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

GROUP B: Patients receive abiraterone acetate PO QD, prednisone PO twice daily (BID), physician's choice ADT, and niraparib PO QD. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 14 days, at 30-90 days, and then every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Completion of informed consent prior to any study specific procedures. Consent may be done remotely.
* Patients must agree to tissue collection for correlative studies at the specified timepoints
* Male aged 18 years and above
* Histologically or cytologically confirmed prostate carcinoma
* Localized or regional high-risk disease as defined by at least one of the following features: Prostate specific antigen (PSA) > 20 ng/mL, T3a or higher, grade group 4-5 (i.e. Gleason score ≥ 8) as per National Comprehensive Cancer Network (NCCN) Prostate Cancer Version 2.2020 for high risk or very high risk prostate cancer, and/or regional lymph nodes positive for prostate cancer
* Planned for definitive treatment of local regional prostate cancer using XRT and androgen ablation
* Willing to undergo ongoing medical castration to maintain testosterone levels of ≤ 50 ng/dL (≤ 2.0 nM) throughout systemic treatment or have undergone bilateral orchiectomy
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2. Patients must have adequate organ and bone marrow function measured within 7 days prior to treatment registration as defined below:
* Hemoglobin ≥ 10.0 g/dL
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
* White blood cells (WBC) > 3 x 10^9/L
* No features suggestive of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) on peripheral blood smear
* Platelet count ≥ 100 x 10^9/L
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (except for patients with known Gilbert's disease). (Note: In subjects with Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤ 1.5 x ULN, subject may be eligible.)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x institutional upper limit of normal
* Calculated creatinine clearance (Cockcroft-Gault Equation) ≥ 30 mL/min
* Serum Albumin ≥ 3.0
* Serum potassium ≥ 3.5 mmol/L
* Able to swallow study drugs whole as a tablet/capsule
* Patients who have partners of childbearing potential (e.g. female that has not been surgically sterilized or who are not amenorrheic for ≥ 12 months) must be willing to use two methods of birth control including adequate barrier protection during the study and for 4 months after last dose of niraparib, abiraterone acetate, and/or apalutamide administration. In addition men should not donate sperm during this period. Please note that the efficacy of hormonal contraception may be decreased if administered with niraparib, abiraterone acetate, and/or apalutamide
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Medications known to lower the seizure threshold must be discontinued or substituted at least 4 weeks prior to study entry

Exclusion Criteria:

* Any prior systemic treatment for prostate cancer with the exception of ADT started within 6 months of trial enrollment. Any prior PARP inhibitor therapy
* Patients who have prostate cancer with distant metastatic disease
* Patients who have had prior major surgery (prostatectomy) or radiotherapy for the treatment of prostate cancer
* Any unresolved toxicity (Common Terminology Criteria for Adverse Events [CTCAE] grade ≥ 2) from previous anti-cancer therapies
* History or current diagnosis of MDS/AML, and/or history of any malignancy [other than the one treated in this study] which has a ≥ 30% probability of recurrence within 24 months (except for adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix or Ta urothelial carcinomas)
* Active uncontrolled infection (patients completing a course of antibiotic or antiviral therapy whose infection is deemed to be controlled may be allowed on study after discussion with the principal investigator [PI]; the PI will serve as the final arbiter regarding eligibility)
* Active or symptomatic viral hepatitis or chronic liver disease
* Active pneumonitis or extensive bilateral lung disease of non-malignant etiology
* Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events. Examples include, but are not limited to superior vena cava syndrome, extensive bilateral lung disease on high resolution computed tomography (HRCT) scan, uncontrolled seizures, history of allogeneic organ transplant, history of primary immunodeficiency or any psychiatric disorder that prohibits obtaining informed consent
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of study medication
* Patients with a known hypersensitivity to niraparib, apalutamide, and/or abiraterone acetate
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness
* Seizure or known condition that may pre-dispose to seizure (e.g. prior stroke within 1year to randomization, brain arteriovenous malformation, Schwannoma, meningioma, or other benign central nervous system [CNS] or meningeal disease which may require treatment with surgery or radiation therapy)
* Severe or unstable angina, myocardial infarction (within 6 months prior to enrollment), symptomatic congestive heart failure, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), uncontrolled hypertension, or clinically significant ventricular arrhythmias within 6 months prior to randomization
* Current evidence of any of the following:

  * Gastrointestinal disorder affecting absorption
  * Active uncontrolled infection (e.g., human immunodeficiency virus [HIV] or viral hepatitis)
  * Any chronic medical condition requiring a higher dose of corticosteroid than 10 mg prednisone/prednisolone once daily
  * Avoid concomitant strong CYP3A4 inducers during abiraterone acetate treatment. If a strong CYP3A4 inducer must be co-administered, increase the abiraterone acetate dosing frequency
  * Avoid co-administration of abiraterone acetate with CYP2D6 substrates that have a narrow therapeutic index. If an alternative treatment cannot be used, exercise caution and consider a dose reduction of the concomitant CYP2D6 substrate
  * Baseline moderate and severe hepatic impairment (Child-Pugh class B & C)
  * Any condition that in the opinion of the investigator, would preclude participation in this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2026-06-07 (Estimated); Study Completion 2026-06-07 (Estimated)

PRIMARY OUTCOMES:
Composite radiographic progression-free survival(rPFS) and biochemical (PSA) progression-free survival (PFS) | From randomization until progression, death, or last assessment without progression, whichever comes first, assessed at 3 years

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Up to 3 years
  Adverse events will be recorded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 along with date and attribution to study treatment.
Incidence and severity of serious adverse events (SAEs) | Up to 3 years
  Graded by NCI CTCAE version 5.0.
Overall survival | From randomization until death or last contact, whichever comes first, assessed up to 3 years
Eugonadal progression-free survival | From randomization until progression, death, or last assessment without progression, whichever comes first, assessed up to 3 years
  Assessed as composite radiographic PFS (rPFS) and biochemical (prostate specific antigen [PSA]) PFS among patients with non-castrate level testosterone. Eugonadal is defined as non-castrate levels of testosterone (> 50 ng/mL).
Progression-free survival | From randomization until progression, death, or last assessment without progression, whichever comes first, assessed up to 3 years
  Defined as composite rPFS and biochemical (PSA) PFS in those with unfavorable histologic response versus favorable histologic response in men who received maximal androgen signaling ablation prior to definitive radiation. PFS will be calculated from histologic response assessment between Parts 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick G Pilie, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org